CLINICAL TRIAL: NCT05240144
Title: Effect of Isometric Handgrip Exercises on Blood Pressure of Hypertensive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sidra Iqbal
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: Blood pressure; Systolic blood pressure; Diastolic blood pressure; Isometric handgrip exercises; Maximal voluntary contraction
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IHG group (Experimental): Isometric handgrip exercises will be performed in 4 sets for 2 min at 30% Maximal Voluntary Contraction (MVC) on both hands with the frequency of 3 days per week for a period of 6 weeks.
  Interventions: Other: IHG
- Aerobic training group (Active Comparator): Aerobic Exercises include walk for 50 min with the frequency of 3 days per week. This exercise will be done for a 6-week period.
  Interventions: Other: Aerobic exercises
- IHG + Aerobic exercises group (Sham Comparator): Isometric handgrip exercises will be performed in 4 sets for 2 min at 30% MVC on both hands with the frequency of 3 days per week for a period of 6 weeks.
  Isometric handgrip exercises will be performed in 4 sets for 2 min at 30% MVC on both hands with the frequency of 3 days per week for a period of 6 weeks.
  Interventions: Other: IHG; Other: Aerobic exercises
- Sham IHG group (Sham Comparator): Isometric handgrip exercises will be performed in 4 sets for 2 min at 5% MVC on both hands with the frequency of 3 days per week for a total 6-week period.
  Interventions: Other: Sham IHG

INTERVENTIONS:
Other: IHG — Isometric handgrip exercises will be performed for 4 x 2 min with the frequency of 3 days per week for a period of 6 weeks.
  Arms: IHG + Aerobic exercises group; IHG group
Other: Aerobic exercises — Aerobic exercise according to the American College of Sports Medicine (ACSM) guidelines that provide the specific criteria as 50 minutes exercises for 3 days a week for a period of 6 weeks.
  Arms: Aerobic training group; IHG + Aerobic exercises group
Other: Sham IHG — Isometric handgrip exercises will be performed in 4 sets for 2 min at 5% MVC on both hands with the frequency of 3 days per week for a total 6-week period
  Arms: Sham IHG group

SUMMARY:
This study is designed to determine the effects of isometric handgrip exercises as compared to aerobic exercises in the hypertensive population, specifically in pre-hypertensives and those with hypertension stage I who are not taking pharmacological treatment. This exercise is designed as part of lifestyle modification for these patients and if proven effective, it can provide an easier to perform exercise regimen as an alternative to be incorporated in the exercise plan of patients who have difficulty in performing aerobic exercises because of musculoskeletal concerns.

DETAILED DESCRIPTION:
Hypertension (HTN) is a significant public health problem, with an increasing worldwide prevalence. The disease has an impact on reducing the quality of life (QOL) and can be life-threatening if not treated early. It is considered the major risk factor for cardiovascular and renal diseases. Complications of hypertension can lead to a variety of serious diseases like stroke, heart attack, and even cardiac and renal failure. Non-pharmacological management via lifestyle modification is focused in the initial stages of HTN through the reduction in alcohol consumption, cessation of tobacco smoking, maintenance of body weight, improvements in nutrition, and increases in physical activity. Physical activity improves health status and prevents the complications of hypertension like stroke and heart failure.

Typically, aerobic exercises in the form of walking and jogging are advised as part of lifestyle modification. effectiveness of resistance training is also worked upon. A relatively newer approach in the form of Isometric Hand Grip exercises (IHG) is also under research because it can serve as a useful alternative for patients who cannot perform aerobic exercises because of musculoskeletal conditions. This study is targeted to assess the effects of IHG exercises, aerobic training, both aerobic and IHG training as well as sham IHG treatment for a comprehensive assessment of effects of IHG training.

ELIGIBILITY:
Inclusion Criteria:

* Pre-hypertension (systolic BP 120-139 mmHg and diastolic BP<80) or stage I hypertensive patients (systolic BP 140-159 mmHg and diastolic BP 90-99mm Hg.

Exclusion Criteria:

* Patients who are taking antihypertensive agents
* Malignant hypertension
* Physical limitation preventing IHG training (e.g., missing arm, severe hand arthritis, carpal tunnel syndrome, or having a musculoskeletal disorder affecting the upper limb.
* Active systemic illness that restricts exercise
* People doing exercise regularly
* Any other cardiopulmonary, metabolic, neurological, or psychiatric illness.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 6 weeks
  Pressure exerted by flowing blood on walls of blood vessels during contraction of heart.
Diastolic blood pressure | 6 weeks
  Pressure exerted by flowing blood on walls of blood vessels during relaxation of heart.
Mean arterial pressure (MAP) | 6 weeks
  Mean arterial pressure (MAP) is the average of arterial pressure during one cardiac cycle and it will be calculated by using the formula MAP = DBP+ 1/3 (SBP-DBP).

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Comprehensive Rehabilitation Center, Bahawalpur, AL, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SH, Chae YR. Characteristics of Aerobic Exercise as Determinants of Blood Pressure Control in Hypertensive Patients: A Systematic Review and Meta-Analysis. J Korean Acad Nurs. 2020 Dec;50(6):740-756. doi: 10.4040/jkan.20169. PMID 33441523
- [Background] Palmeira AC, Farah BQ, Silva GOD, Moreira SR, Barros MVG, Correia MA, Cucato GG, Ritti-Dias RM. Effects of isometric handgrip training on blood pressure among hypertensive patients seen within public primary healthcare: a randomized controlled trial. Sao Paulo Med J. 2021 Nov 15;139(6):648-656. doi: 10.1590/1516-3180.2020.0796.R1.22042021. eCollection 2021. PMID 34787298
- [Background] Shafi ST, Shafi T. A survey of hypertension prevalence, awareness, treatment, and control in health screening camps of rural central Punjab, Pakistan. J Epidemiol Glob Health. 2017 Jun;7(2):135-140. doi: 10.1016/j.jegh.2017.01.001. Epub 2017 Feb 8. PMID 28188121
- [Background] Silva GO, Farah BQ, Germano-Soares AH, Andrade-Lima A, Santana FS, Rodrigues SL, Ritti-Dias RM. Acute blood pressure responses after different isometric handgrip protocols in hypertensive patients. Clinics (Sao Paulo). 2018 Oct 18;73:e373. doi: 10.6061/clinics/2018/e373. PMID 30365821
- [Background] Farah BQ, Germano-Soares AH, Rodrigues SLC, Santos CX, Barbosa SS, Vianna LC, Cornelissen VA, Ritti-Dias RM. Acute and Chronic Effects of Isometric Handgrip Exercise on Cardiovascular Variables in Hypertensive Patients: A Systematic Review. Sports (Basel). 2017 Aug 1;5(3):55. doi: 10.3390/sports5030055. PMID 29910415
- [Background] Herrod PJJ, Doleman B, Blackwell JEM, O'Boyle F, Williams JP, Lund JN, Phillips BE. Exercise and other nonpharmacological strategies to reduce blood pressure in older adults: a systematic review and meta-analysis. J Am Soc Hypertens. 2018 Apr;12(4):248-267. doi: 10.1016/j.jash.2018.01.008. Epub 2018 Feb 2. PMID 29496468